CLINICAL TRIAL: NCT02514876
Title: Visualization of Human Cardiovascular Anatomy With Foresight Intracardiac Echocardiography (ICE) System
Brief Title: Foresight Intracardiac Echocardiography (ICE) System
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Conavi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: EXT-001
Record Dates: First submitted 2015-07-27; First posted 2015-08-04 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

ARMS (1):
- Single arm- Foresight ICE System (Experimental): This open label feasibility study will evaluate the Foresight ICE system for imaging chambers of the heart and guiding transseptal puncture during an atrial fibrillation (AF) ablation procedure.
  Interventions: Device: Foresight ICE System

INTERVENTIONS:
Device: Foresight ICE System — The Foresight ICE System is composed of a sterile, single-use catheter intended to operate with a Foresight ICE PIM and Hummingbird Console.

SUMMARY:
This study will evaluate the efficacy of 2D forward-looking and 3D Intracardiac Echocardiography (ICE) to guide septal punctures during Atrial Fibrillation ablation procedures.

DETAILED DESCRIPTION:
This study is part of a multiphase study. Phase 1 involves 10 patients at a single centre. Phase 2 will be done a multi centre study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years old.
* Patient is undergoing an atrial fibrillation ablation procedure.
* Patient has a transesophageal echocardiogram (TEE) within the 48 hours prior to ablation procedure to rule out left atrial thrombus.
* Patient provides informed, written consent for participation in the study.

Exclusion Criteria:

* Patients in whom placement of an ICE catheter in the right atrium for adequate atrial visualization is not technically feasible (as evaluated and determined by the physician performing the procedure).
* Patients in whom transseptal puncture is relatively contraindicated.
* Patients in whom left atrial clot or dense spontaneous contrast is identified on TEE, which would increase thromboembolic risk.
* Women of child bearing potential, in whom pregnancy cannot be excluded.
* Patients unable to grant informed, written consent for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04-08 (Actual); Study Completion 2016-05-05 (Actual)

PRIMARY OUTCOMES:
Successful transseptal puncture during atrial fibrillation ablation procedure under the guidance of study device | During ablation procedure (2-4 h)

CONTACTS AND LOCATIONS:
Overall Officials: Atul Verma, MD, Principal Investigator — Southlake Regional Health Centre
Locations (1):
- Southlake Regional Health Centre, Newmarket, Ontario, Canada